CLINICAL TRIAL: NCT06983327
Title: Brief Intervention for Chronic Pain and History of Stressful Experiences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Robert Edwards, Clinical Psychologist, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024P001483
Record Dates: First submitted 2025-04-14; First posted 2025-05-21 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Chronic Pain; Trauma; Adverse Childhood Experiences
MeSH Terms: conditions — Chronic Pain; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brief Intervention (Experimental)
  Interventions: Behavioral: Trauma Focused Emotional Awareness and Expression Therapy (EAET)

INTERVENTIONS:
Behavioral: Trauma Focused Emotional Awareness and Expression Therapy (EAET) — The intervention is three-session program which includes pain neuroscience education, education on the relationship between trauma and chronic pain, and skills training to reduce pain- and stress-related symptoms.

SUMMARY:
The goal of this study is to understand whether a brief, three session program can be helpful in reducing symptoms related to both chronic pain and stressful experiences/trauma.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a chronic pain condition (pain for at least 3 months or more)
* History of psychosocial trauma or stressful experience (Adverse Childhood Events questionnaire [ACEs] score of ≥ 3 OR Trauma History Questionnaire Score [THQ] of ≥ 2)
* English fluency
* Access to a smartphone, laptop, or computer
* Able to participate in the intervention via a virtual platform

Exclusion Criteria:

* Unable to participate in 3 weekly sessions
* Unable to complete study procedures due to the presence of delirium, dementia, psychosis, or other cognitive impairment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-02-14 (Actual); Primary Completion 2025-11-28 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of Recruitment | At screening
  Feasibility of recruitment: Rate of ≥70% of the patients who are identified as eligible for the study will agree to participate and enroll.
Treatment Completion | From enrollment to end of treatment at 4 weeks
  Rate of ≥70% of participants who start the intervention will complete at least 2 of the 3 sessions.
Feasibility of Data Collection | At end of treatment at (~4 weeks post-enrollment), and at 1-month follow-up (~8 weeks post-enrollment)
  Rate of ≥70% of participants will complete the survey at end of treatment and at 1-month follow-up.
Treatment Credibility | At end of treatment at (~4 weeks post-enrollment), and at 1-month follow-up (~8 weeks post-enrollment)
  Rate of ≥70% of participants will report average credibility and expectancy scores greater than the scale's midpoint.
Treatment Helpfulness | At end of treatment at (~4 weeks post-enrollment), and at 1-month follow-up (~8 weeks post-enrollment)
  Rate of ≥70% participants will report average treatment helpfulness scores greater than the scale's midpoint.

SECONDARY OUTCOMES:
Pain Interference | At end of treatment at (~4 weeks post-enrollment), and at 1-month follow-up (~8 weeks post-enrollment)
  Pain interference Sub-scale of the Patient-Reported Outcomes Measurement Information System-29 (PROMIS-29). Range 4-20; higher scores indicate worse pain interference.
Pain Catastrophizing | At end of treatment at (~4 weeks post-enrollment), and at 1-month follow-up (~8 weeks post-enrollment)
  Pain Catastrophizing Scale (PCS); Range 0-52; higher scores indicate worse pain catastrophizing.
Posttraumtic Stress Disorder (PTSD) Symptoms | At end of treatment at (~4 weeks post-enrollment), and at 1-month follow-up (~8 weeks post-enrollment)
  PTSD Checklist for DSM-5 (PCL-5); Range 0-80; higher scores indicate worse PTSD symptoms.
Kinesiophobia | At end of treatment at (~4 weeks post-enrollment), and at 1-month follow-up (~8 weeks post-enrollment)
  Tampa Scale of Kinesiophobia (TSK); Range 17-68; higher scores indicate worse kinesiophobia.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Chestnut Hill, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No